CLINICAL TRIAL: NCT00341835
Title: Genetic Epidemiology of Lung Cancer
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903288; 03-HG-N288
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer
Keywords: Association; Genetics; Linkage
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High risk lung cancer families: Individuals from families with a high risk of lung cancer, both affected and unaffected family members

SUMMARY:
This study will search for genes that greatly increase the risk of developing lung cancer in conjunction with cigarette smoking or other environmental agents, or both. Lung cancer is the second most common cancer diagnosed among men and women and the leading cause of cancer death in the United States. It has been frequently given as an example of cancer determined only by the environment, certain occupations, and dietary habits. Yet researchers have long had a hypothesis that people vary in their risk of becoming affected when exposed to these factors. Also, some evidence has shown that lung cancer in families may be due to the combined effects of inheritance of a major gene and cigarette smoking.

Individuals who have a confirmed diagnosis of lung cancer or a family history of lung cancer may be eligible to enroll their families in the study.

Family members will be asked to do one or more of the following:

* Complete a questionnaire about personal medical history, lifestyle, and diet.
* Have blood drawn from a vein in the arm.
* If a family member has had a biopsy or is scheduled for one, give permission to obtain medical records and a portion of the stored tissue.
* If any relatives have died of cancer, sign a release form to allow researchers to get copies of medical and pathology records, and tissue samples from surgery.

If the family members agree, they may be recontacted to answer questions about their health and those of their family, during an annual telephone conversation. Follow-up questionnaires may be sent to participants, to determine if any new cancers have developed in the family. In the event of a new cancer, the classification of the family may change from the low-risk to intermediate risk-level and from the intermediate-risk to high-risk level. Follow-up will continue, to get information about tumors and death. Also, a newsletter for lung cancer families will occasionally be distributed to participants. In the future, the Internet will also provide information for families.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in the US, and represents a significant burden on health care resources. Accumulated evidence suggests that there are genetic susceptibility components in lung cancer, and that gene-environment interactions are important. While major breakthroughs have been made in understanding the genetic susceptibility basis of other cancers, studies to identify specific major loci affection lung cancer risk are notably lacking. The high case fatality rate (14 percent 5-year survival rate) and low resection rate (25 percent) makes the study of lung cancer families particularly challenging because it is difficult to collect adequate numbers of biospecimens for DNA analysis. Only a collaborative effort to identify, accrue, and genotype familial lung cancer (FLC) families will be successful in characterizing the genetic basis of familial lung cancer.

This project is part of a multi-center, multi-investigator, interdisciplinary team highly experienced in genetic epidemiology, gene mapping, lung biology, and cancer molecular genetics, known as the Genetic Epidemiology of Lung Cancer Consortium (GELCC) formed to identify a lung cancer susceptibility gene(s) and to estimate gene-environment interaction in the etiology of this neoplasm in order to elucidate a strategy for the prevention, control and clinical management of this disease through identification of genetically high-risk individuals.

Confirmation of a genetic predisposition for lung cancer may be possible by using linkage analysis to localize the putative susceptibility gene to a specific chromosomal region. The strength of linkage analysis is dependent upon the recruitment of multiple large kindreds for which tissue samples are available and the history of tumor incidence exists for two, preferably more, generations. Our strategy is to combine the most informative pedigrees but preferably eventually up to 500 pedigrees. This strategy yields a substantial increase in power and cost-effectiveness over the usual strategy of each site working independently and genotyping many marginally informative families. To date this strategy appears successful, in that results from our first 52 genotyped families resulted in significant evidence in favor of linkage to a region on chromosome 6q and suggestive evidence for several other regions. We believe that ongoing data collection and analysis of these preliminary results will also be fruitful. Recently, the National Cancer Institute funded this ongoing project in a competitive renewal (5 years) of our multi-center R01 that supports data collection and work at all sites besides NHGRI and NCI.

All data collection is under the direction of each P.I. at the data collection sites and funded by their respective grants and contracts. NHGRI investigators do not have any contact with study subjects and no NHGRI employees receive any funds from these grants. Because this disorder is complex and has a high likelihood of being caused by multiple loci, multiple parametric and non-parametric methods of analysis will be employed. Heterogeneity will be taken into account during these analyses, as will environmental covariates, such as the effect of smoking. Only statistical analyses are performed at the NHGRI site, but laboratory work ranging from genotyping, sequencing, array CGH, model organism experiments and other methods occurs at other sites as part of this collaboration.

ELIGIBILITY:
* INCLUSION CRITERIA:

All individuals with a histologically confirmed diagnosis of lung cancer or a family of lung cancer are eligible to enroll their family in the study. Five major histologic types of lung cancer, i.e., adenocardinoma, squamous cell, small cell, large cell, and unspecified nonsmall cell carcinoma will be included. In addition to lung cancer patients, LSU will also contact patients newly diagnosed with bronchus or tracheal cancer in target hospital areas to request their enrollment in their study. In addition, several sites including LSU, Mayo Clinic and Karmanos Cancer Institute also collect DNA samples from unaffected, geographically and ethnically matched controls.

For the purposes of this study, an eligible family must meet the minimum criteria for familial lung cancer: at least 2 first-degree relatives in the family have had lung cancer. Priority will be given to more highly loaded pedigrees and to families in which the affected persons had onset of the disease at an early age (less than 50 years). Lung cancer cases may be living or deceased. Relatives with lung cancer are defined as first- o second-degree relatives or cousins of index cases will be eligible to participate in the study because their familial relationships might provide useful linkage information.

Adult participants must be physically able to tolerate removal of 25 to 40 ml of blood, or buccal brush sampling of their cheek. Children above 5 years old must be able to physically tolerate an amount of blood drawn that is equal to 4ml/kg of their weight. Adults must be willing to complete a self-administered environmental exposure questionnaire, and all participants must be able to consent to the study procedures (or have appropriate assent/parental consent). Biological specimens, including blood samples, archived tumor blocks and other medical records will be obtained from patients treated at the various hospitals and collection sites and from individuals with strong family history of lung cancer (either affected or unaffected) who have either been self-referred or physician referred to the study.

EXCLUSION CRITERIA:

Excluded from the study are families or individuals within the family who do not meet the minimum criteria described above. Individuals who do not sign the Consent Form will be excluded, and families for whom all necessary members do not sign the Consent Form may be excluded. MAYO also excludes patients who (1) do not speak English, (2) are non-US citizens or residents and (3) are diagnosed with an uncommon tumor type that is not among the above specified types (e.g.) mixed cell or unspecified non-small cell lung cancer, carcinoids, sarcomas and lymphomas of the lung and bronchus). This is done at MAYO because the family study is piggy-backed onto a case-control study. No fetuses, prisoners or institutionalized individuals will be enrolled. While this study does not target pregnant women, because contact with many of the families will be by mail we will not be able to exclude pregnant women. Additionally, the participant's own physician or health care clinic will draw blood samples from long-distance participants and therefore can determine if there is any risk to the woman or her fetus. UMHS also excludes children as research participants in their site.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: These are coded samples and data that were previously collected at multiple clinical data collection sites. They were mainly identified through a clinical site that diagnosed one family member with lung cancer and then offered enrollment in this study because of additional family history of disease. No study participants are enrolled at the NIH.@@@
Sampling Method: Non-Probability Sample
Enrollment: 6356 (Actual)
Dates: Start 2003-08-26 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Determine whether there are genetic variants contributing to lung cancer risk | ongoing
  Determine whether there are genetic variants contributing to lung cancer risk

SECONDARY OUTCOMES:
Determine whether there are gene-gene or gene-environment interactions contributing to lung cancer risk | ongoing
  Determine whether there are gene-gene or gene-environment interactions contributing to lung cancer risk

CONTACTS AND LOCATIONS:
Overall Officials: Joan Bailey-Wilson, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States